CLINICAL TRIAL: NCT06523361
Title: Contribution of Immersive Virtual Reality to a Standardized Rehabilitation Program for Upper Limb Chronic Pain: A Single-Case Experimental Design Study
Acronym: ReVIDoC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 49RC24_0066
Record Dates: First submitted 2024-07-04; First posted 2024-07-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Complex Regional Pain Syndrome Type I of the Upper Limb
MeSH Terms: conditions — Reflex Sympathetic Dystrophy

STUDY DESIGN:
Intervention Model Description: Single case experimental design, with sequential introduction of the intervention and comparison within subject (between phases) and between subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- introduction of the intervention phase before session 4 with occupational therapist (Other): The first "group" will be repeated three times. For each participant, the beginning of the intervention will be randomized. All participants will undergo a baseline phase, intervention phase, and follow-up phase. During the baseline phase, participants serve as controls. As the randomized beginning of the intervention varies across subjects, the length of the baseline phase also varies. The objective is to identify a change in the outcome measure when the intervention starts, despite the differing lengths of the baseline phases across participants.
  Interventions: Device: H'ability
- introduction of the intervention phase before session 5 with occupational therapist (Other): The second "group" will be repeated three times. For each participant, the beginning of the intervention will be randomized. All participants will undergo a baseline phase, intervention phase, and follow-up phase. During the baseline phase, participants serve as controls. As the randomized beginning of the intervention varies across subjects, the length of the baseline phase also varies. The objective is to identify a change in the outcome measure when the intervention starts, despite the differing lengths of the baseline phases across participants.
  Interventions: Device: H'ability
- introduction of the intervention phase before session 6 with occupational therapist (Other): The third "group" will be repeated three times. For each participant, the beginning of the intervention will be randomized. All participants will undergo a baseline phase, intervention phase, and follow-up phase. During the baseline phase, participants serve as controls. As the randomized beginning of the intervention varies across subjects, the length of the baseline phase also varies. The objective is to identify a change in the outcome measure when the intervention starts, despite the differing lengths of the baseline phases across participants.
  Interventions: Device: H'ability
- introduction of the intervention phase before session 7 with occupational therapist (Other): The fourth "group" will be repeated three times. For each participant, the beginning of the intervention will be randomized. All participants will undergo a baseline phase, intervention phase, and follow-up phase. During the baseline phase, participants serve as controls. As the randomized beginning of the intervention varies across subjects, the length of the baseline phase also varies. The objective is to identify a change in the outcome measure when the intervention starts, despite the differing lengths of the baseline phases across participants.
  Interventions: Device: H'ability

INTERVENTIONS:
Device: H'ability — H'ability is introduced depending the randomization result, during the baseline (before session 4, 5, 6 or 7 with occupational therapist

SUMMARY:
Background: Chronic pain represents a significant public health concern, given its high prevalence and the substantial impact it has on the quality of life of many individuals affected. There is no single, universally effective medical treatment for chronic pain. The gold standard for treatment is a multidisciplinary rehabilitation program. Immersive virtual reality (IVR) represents a novel and promising approach to do rehabilitation, offering the potential to enhance engagement and perception of movement.

The objective of this study was to investigate the improvement of upper limb function in chronic pain patients using an IVR device in occupational therapy sessions during a rehabilitation program.

Methods: The study use a single-case experimental design (SCED) to investigate the efficacy of IVR device in improving upper limb function in patients with upper limb chronic pain. The study was conducted in three phases: baseline, intervention, and follow-up. The SCED will be with multiple baseline across subjects, whereby the patient serves as his own control. A total of 12 participants will be included. The virtual reality sessions will be conducted exclusively during the intervention phase. The primary outcome measure will be the upper limb function, as assessed by the Quick DASH (Disabilities of the Arm, Shoulder and Hand) questionnaire. Furthermore, the intensity of pain will be quantified using a numeric scale, and the pain self-efficacy will be evaluated using the Pain Self-Effacity Short Form Questionnaire.

Expected results: This method will allow for the comparison of phases within and between subjects to determine whether the IVR sessions improve the function assessed by the Quick DASH.

Conclusion: Further investigation is required to determine the potential benefits of using IVR for upper limb chronic pain rehabilitation, with a particular focus on the development of precise protocols for its use in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain in the upper limb, predominantly in one or both upper limbs, for more than 3 months
* Age between 18 and 65
* Patient affiliated with or benefiting from a social security organization
* Person able to tolerate the virtual reality device
* Informed consent form signed

Exclusion Criteria:

* Upper limb surgery < 6 months
* Infection or pathology of the central nervous system or active cancer
* Fibromyalgia
* Severe psychiatric or cognitive disorders
* Diabetes mellitus complicated by peripheral neuropathy
* Neurogenic paraosteoarthropathy or recent fracture
* Pregnancy or breast-feeding.
* Poor understanding of the French language.
* Person deprived of liberty by judicial or administrative decision
* Psychiatric disorder
* Person subject to a legal protection measure
* Person unable to give consent
* In connection with the virtual reality device: unstabilized epilepsy, facial trauma < 3 months, hearing or visual impairment, pain, dizziness or nausea caused by the use of virtual reality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Quick DASH (Quick Disabilities of the Arm, Shoulder and Hand) self-questionnaire | 5 times per week for 7 weeks
  The self-questionnaire contains 11 items to assess the patient's ability to perform certain activities of daily living, the severity of the pain, the impact of the condition on social or professional life, etc. rated on a scale of 1 (no difficulty or inability) to 5 (unable to do)

SECONDARY OUTCOMES:
self-assessment of pain using the Numerical Scale (EN) | 5 times per week for 7 weeks
  numerical scale from 1 to 10
subjective assessment of pain via the PSEQ-2 self-questionnaire | 5 times per week for 7 weeks
  PSEQ-2 (Pain Self Efficacy Questionnaire). measure patients' confidence in their ability to perform tasks despite pain-scale from 0 to 6.
functional assessment of the shoulder using the C-test | 5 times per week for 7 weeks
  measurement of the thoracohumeral angle during active elbow elevation
self-evaluation of performance and feeling of satisfaction associated with the difficulties identified by the patient with MCRO questionnaire | One time between day 7 and day 14 + one time between week 6 and week 7.
  Mesure Canadienne du Rendement Occupationnel (MCRO). Scale from 1 to 10
Measure of Constant score:composite score allowing to assess pain, level of daily activities, level of hand work, shoulder mobility and strength. | One time between day 7 and day 14 + one time between week 6 and week 7.
  composite score allowing to assess pain, level of daily activities, level of hand work, shoulder mobility and strength.
assessment of kinesiophobia with the Tampa Scale for Kinesiophobia (TSK) | once at inclusion + one time between week 6 and week 7.
  reliable and validated self-questionnaire in French which assesses through 17 items the fear of movement in connection with the fear of being injured during a movement (25). Each question is scored between 1 (strongly disagree) and 4 (strongly agree) with the exception of items 4, 8, 12 and 16 which are inversely scored with 1 (strongly agree ) and 4 (strongly disagree). A total score greater than or equal to 40 confirms significant kinesiophobia and the higher the score, the greater the kinesiophobia.
assessing grip strength with the Jamar test | One time between day 7 and day 14 + one time between week 6 and week 7.
  This is a quick and simple test that requires squeezing a hydraulic dynanometer to its fullest extent. 3 repeated measurements are taken on one side then the other and only the highest value is retained for each side. It has been shown in the literature that grip strength is a good indicator of overall upper limb strength and that muscle strength in a chronically painful limb is reduced.
assessing dexterity with the Box and Block Test (BBT) | One time between day 7 and day 14 + one time between week 6 and week 7.
  It consists of 150 cubes placed in a wooden box with two equal-sized compartments. The patient must move, with one hand, a maximum of cubes from one compartment to another, one by one, in 1 minute. The score obtained corresponds to the number of cubes moved for each hand in one minute.
assessing dexterity with the Purdue Pegboard Test (PPT) | One time between day 7 and day 14 + one time between week 6 and week 7.
  The test involves taking small metal pegs and placing them in the small holes of a standardized board for 30 seconds
self-assessment of the H'ability© device according to healthcare professionals and patients using the SUS scale (System Usability Scale) | one time between week 6 anD week 7.
  questionnaire for measuring the usability of interactive systems, validated in French, which includes 10 items associated with a 5-point Likert scale (from 1 = Completely disagree to 5 = Completely agree). The overall score is obtained by subtracting 1 from the score checked for items 1, 3, 5, 7 and 9, then calculating 5 minus the score checked for items 2, 4, 6, 8 and 10 (items whose wording is negative and reverse rating). The 10 scores thus calculated are added and multiplied by 2.5, to obtain a total score between 0 and 100 (a higher score means better usability).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Angers, Angers
  - CH LAVAL, Laval